CLINICAL TRIAL: NCT00598676
Title: Intracoronary Stenting and Angiographic Results: Test Efficacy of 3 Limus-Eluting STents (ISAR-TEST 4): Prospective, Randomized Trial of 3-limus Agent-eluting Stents With Different Polymer Coatings
Brief Title: 3 Limus Agent Eluting Stents With Different Polymer Coating
Acronym: ISAR-TEST-4
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Prof. A. Schömig, Deutsches Herzzentrum Munich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GE IDE No. S02607
Record Dates: First submitted 2008-01-10; First posted 2008-01-22 (Estimated); Last update posted 2010-03-15 (Estimated); Status verified 2010-03

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- BPRES (Experimental): biodegradable polymer rapamycin-eluting stent
  Interventions: Device: biodegradable polymer Rapamycin-eluting stent
- PPRES (Active Comparator): permanent polymer rapamycin-eluting stent
  Interventions: Device: permanent polymer rapamycin-eluting stent (Cypher)
- PPEES (Active Comparator): permanent polymer everolimus-eluting stent
  Interventions: Device: permanent polymer everolimus-eluting stent (Xience, Promus)

INTERVENTIONS:
Device: biodegradable polymer Rapamycin-eluting stent — due to randomization, rapamycin-eluting stent with biodegradable polymer will be implanted
  Other Names: ISAR stent
  Arms: BPRES
Device: permanent polymer rapamycin-eluting stent (Cypher) — due to randomization, rapamycin-eluting stent with permanent polymer will be implanted
  Other Names: Cypher
  Arms: PPRES
Device: permanent polymer everolimus-eluting stent (Xience, Promus) — due to randomization, everolimus-eluting stent with permanent polymer will be implanted
  Other Names: Xience; Promus
  Arms: PPEES

SUMMARY:
The aim of this study is to determine whether biodegradable polymer based rapamycin-eluting stent performs equal to permanent polymer based everolimus- and rapamycin-eluting stents regarding reduction of adverse cardiac events at one year.

DETAILED DESCRIPTION:
Drug-eluting stents significantly reduce in-stent restenosis and the subsequent need for target vessel revascularisation compared with bare metal stents. Although this applies to the vast majority of patients, intimal hyperplasia and in-stent restenosis have not been completely eliminated and remain to occur in certain high risk subgroups. Thus there is ongoing research for new, potentially more effective and safe drug-eluting stent systems.

One direction of extensive research is the search of new polymers such as biodegradable polymers which allow a controlled drug-release and disappear with time, reducing the probability of polymer-induced chronic inflammation on the vessel wall.

Another direction is finding new drugs to suppress neointimal hyperplasia. Promising preclinical and clinical results suggest that the Everolimus eluting stent platform might provide potential improvements over prior generations of drug-eluting stents.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than age 18 with ischemic symptoms or evidence of myocardial ischemia in the presence of ≥ 50% de novo stenosis located in native coronary vessels.
* Written, informed consent by the patient or her/his legally-authorized representative for participation in the study.
* In women with childbearing potential a negative pregnancy test is mandatory

Exclusion Criteria:

* Target lesion located in the left main trunk.
* Target lesion located in the bypass graft.
* In-stent restenosis.
* Cardiogenic shock.
* Malignancies or other comorbid conditions (for example severe liver, renal and pancreatic disease) with life expectancy less than 12 months or that may result in protocol non-compliance.
* Known allergy to the study medications: Clopidogrel, Rapamycin, Everolimus, stainless steel or cobalt chrome.
* Inability to take clopidogrel for at least 6 months.
* Pregnancy (present, suspected or planned) or positive pregnancy test.
* Previous enrollment in this trial.
* Patient's inability to fully cooperate with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2600 (Actual)
Dates: Start 2007-09; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
The primary end point of the study is a combined endpoint of cardiac death, myocardial infarction related to the target vessel or revascularization related to the target lesion. | 12 months

SECONDARY OUTCOMES:
In-segment binary restenosis at follow-up angiography | 6-8 months
Late Lumen Loss at follow-up angiography | 6-8 months
All cause mortality. | 12 months
Incidence of stent thrombosis (by ARC definition) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Albert Schoemig, MD, Study Chair — Deutsches Herzzentrum Muenchen; Adnan Kastrati, MD, Principal Investigator — Deutsches Herzzentrum Muenchen
Locations (2):
- Germany (2):
  - Deutsches Herzzentrum Muenchen, Munich
  - Medizinische Klinik, Klinikum rechts der Isar, München

REFERENCES:
- [Result] Byrne RA, Kastrati A, Kufner S, Massberg S, Birkmeier KA, Laugwitz KL, Schulz S, Pache J, Fusaro M, Seyfarth M, Schomig A, Mehilli J; Intracoronary Stenting and Angiographic Results: Test Efficacy of 3 Limus-Eluting Stents (ISAR-TEST-4) Investigators. Randomized, non-inferiority trial of three limus agent-eluting stents with different polymer coatings: the Intracoronary Stenting and Angiographic Results: Test Efficacy of 3 Limus-Eluting Stents (ISAR-TEST-4) Trial. Eur Heart J. 2009 Oct;30(20):2441-9. doi: 10.1093/eurheartj/ehp352. Epub 2009 Aug 30. PMID 19720642
- [Derived] Coughlan JJ, Aytekin A, Xhepa E, Cassese S, Joner M, Koch T, Wiebe J, Lenz T, Rheude T, Pellegrini C, Gewalt S, Ibrahim T, Laugwitz KL, Schunkert H, Kastrati A, Kufner S. Target and non-target vessel related events at 10 years post percutaneous coronary intervention. Clin Res Cardiol. 2022 Jul;111(7):787-794. doi: 10.1007/s00392-022-01986-4. Epub 2022 Feb 11. PMID 35147767
- [Derived] Lenz T, Koch T, Joner M, Xhepa E, Wiebe J, Coughlan JJ, Aytekin A, Ibrahim T, Fusaro M, Cassese S, Laugwitz KL, Schunkert H, Kastrati A, Kufner S; ISAR-TEST 4 (Intracoronary Stenting, Angiographic Results: Test Efficacy of 3 Limus-Eluting Stents) Investigators dagger. Ten-Year Clinical Outcomes of Biodegradable Versus Durable Polymer New-Generation Drug-Eluting Stent in Patients With Coronary Artery Disease With and Without Diabetes Mellitus. J Am Heart Assoc. 2021 Jun 15;10(12):e020165. doi: 10.1161/JAHA.120.020165. Epub 2021 Jun 2. PMID 34075784
- [Derived] Kufner S, Joner M, Thannheimer A, Hoppmann P, Ibrahim T, Mayer K, Cassese S, Laugwitz KL, Schunkert H, Kastrati A, Byrne RA; ISAR-TEST 4 (Intracoronary Stenting and Angiographic Results: Test Efficacy of 3 Limus-Eluting Stents) Investigators. Ten-Year Clinical Outcomes From a Trial of Three Limus-Eluting Stents With Different Polymer Coatings in Patients With Coronary Artery Disease. Circulation. 2019 Jan 15;139(3):325-333. doi: 10.1161/CIRCULATIONAHA.118.038065. PMID 30586724
- [Derived] Kufner S, Byrne RA, Valeskini M, Schulz S, Ibrahim T, Hoppmann P, Schneider S, Laugwitz KL, Schunkert H, Kastrati A; Intracoronary Stenting and Angiographic Results: Test Efficacy of 3 Limus-Eluting Stents (ISAR-TEST4) Investigators. Five-year outcomes from a trial of three limus-eluting stents with different polymer coatings in patients with coronary artery disease: final results from the ISAR-TEST 4 randomised trial. EuroIntervention. 2016 Mar;11(12):1372-9. doi: 10.4244/EIJY14M11_02. PMID 25405657
- [Derived] Byrne RA, Kastrati A, Massberg S, Wieczorek A, Laugwitz KL, Hadamitzky M, Schulz S, Pache J, Fusaro M, Hausleiter J, Schomig A, Mehilli J; ISAR-TEST 4 Investigators. Biodegradable polymer versus permanent polymer drug-eluting stents and everolimus- versus sirolimus-eluting stents in patients with coronary artery disease: 3-year outcomes from a randomized clinical trial. J Am Coll Cardiol. 2011 Sep 20;58(13):1325-31. doi: 10.1016/j.jacc.2011.06.027. PMID 21920260
- [Derived] Kufner S, Massberg S, Dommasch M, Byrne RA, Tiroch K, Ranftl S, Fusaro M, Schomig A, Kastrati A, Mehilli J; Intracoronary Stenting and Angiographic Results: Test Efficacy of 3 Limus-Eluting Stents Trial Investigators. Angiographic outcomes with biodegradable polymer and permanent polymer drug-eluting stents. Catheter Cardiovasc Interv. 2011 Aug 1;78(2):161-6. doi: 10.1002/ccd.22823. Epub 2011 Mar 11. PMID 21400652